CLINICAL TRIAL: NCT06643182
Title: Effect of Back Support on Vital Signs and Comfort After Transfemoral Angiography
Brief Title: Use of Back Support After Transfemoral Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, associate proffesor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/5744
Record Dates: First submitted 2024-08-13; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-08

CONDITIONS: Patient Engagement; Femoral Angiography
Keywords: femoral angiography; back support; vital signs; comfort
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Back Gupport Group (Experimental): After the transfemoral angiography procedure, the patient will be taken to bed and monitored. Approximately 2 hours after the procedure, under the control of the doctor and nurse, the sheath in the patient's groin area will be pulled and a 3 kg sandbag will be left. A 36x33x10 cm gel-containing visco pillow will be placed in the patient's lumbar cavity by the research nurse and primary nurse to fill the anatomical space. The patient will be monitored in a supine position with the head elevated (30 degrees) and blood pressure, pulse, respiratory rate, oxygen saturation and comfort and pain level will be recorded at 0, 3 and 6 hours.
  Interventions: Other: Back Support
- Control Group (No Intervention): The patients in this group will be monitored in the supine position with the head elevated (30 degrees) without pillow support and blood pressure, pulse, respiratory rate, oxygen saturation and comfort and pain level will be recorded at 0, 3 and 6 hours.

INTERVENTIONS:
Other: Back Support — When the sandbag is to be left by the researcher together with the nurse caring for the patient, the patient will be placed in the left lateral position for a short time, a gel-filled orthopedic non-sweating viscose pillow will be placed in the patient's lumbar region and the patient will be placed in a supine position with the head supported.
  Arms: Back Gupport Group

SUMMARY:
In the routine treatment procedure after coronary angiography (CAG), the patients remain in the supine position for a long time, which leads to decreased venous return and back pain. In addition, lying in the same position for 2 hours or more in the back area causes an increase in pressure. Increased pressure disrupts cell and tissue blood supply. The resulting pain may increase sympathetic stimulation. Therefore, sympathetic stimulation increases heart rate, blood pressure, myocardial oxygen consumption and cardiac workload. After the transfemoral coronary angiography (CAG) procedure, which is frequently applied to adults for both diagnosis and treatment, the back support to be applied to ensure that the vital signs (pulse, blood pressure, respiratory rate and blood oxygen saturation) of the patients remain stable and to increase their comfort level can prevent the deviation of the vital signs of the patients from normal and contribute to the treatment process with patient satisfaction.

DETAILED DESCRIPTION:
In the routine treatment procedure after coronary angiography (CAG), the patients remain in the supine position for a long time, which leads to decreased venous return and back pain. In addition, lying in the same position for 2 hours or more in the back area causes an increase in pressure. Increased pressure disrupts cell and tissue blood supply. The resulting pain may increase sympathetic stimulation. Therefore, sympathetic stimulation increases heart rate, blood pressure, myocardial oxygen consumption and cardiac workload. After the transfemoral coronary angiography (CAG) procedure, which is frequently applied to adults for both diagnosis and treatment, the back support to be applied to ensure that the vital signs (pulse, blood pressure, respiratory rate and blood oxygen saturation) of the patients remain stable and to increase their comfort level can prevent the deviation of the vital signs of the patients from normal and contribute to the treatment process with patient satisfaction.

This study will be conducted to evaluate the effect of back support on patients undergoing transfemoral angiography on the patients' vital signs, which are defined as pulse, blood pressure, respiratory rate and blood oxygen saturation (SPO2), as well as comfort levels indicating satisfaction levels.

The study is planned to be completed between September 1, 2024 and April 1, 2025. The universe of the study, which was conducted as a randomized controlled trial model, consisted of patients who underwent angiography in the cardiovascular surgery intensive care units of Tunceli State Hospital. Randomization of the participants was planned to be assigned to the experimental and control groups via random.org (Back support group=40, Control group=40). "Patient Information Form", "Visual Analog Scale (VAS)" and "Immobilization Comfort Scale (IMC)" will be used in data collection. General linear model and mixed ANOVA analysis will be performed according to the characteristics of the data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 who underwent femoral coronary angiography,
* Patients who did not have verbal communication problems,
* Patients who consented to participate in the study were determined as patients.

Exclusion Criteria:

* Patients who underwent radial angiography,
* Have chronic low back pain,
* Have had previous back surgery/herniated disc,
* Have coagulation problems (PLT<50000 mm3),
* Did not consent to participate in the study,
* Have communication problems.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of back support use on pulse | 6 hour (Data collection time for each patient)
  Patients will be monitored for 6 hours in a supported supine position and Pulse will be recorded at 3-hour intervals.
Effect of back support use on blood pressure | 6 hour (Data collection time for each patient)
  Patients will be monitored for 6 hours in a supported supine position and blood pressure will be recorded at 3-hour intervals.m
Effect of back support use on respiratory rate | 6 hour (Data collection time for each patient)
  Patients will be monitored for 6 hours in a supported supine position and respiratory rate will be recorded at 3-hour intervals.m
Effect of back support use on partial oxygen saturation | 6 hour (Data collection time for each patient)
  Patients will be monitored for 6 hours in a supported supine position and partial oxygen saturation will be recorded at 3-hour intervals.m
Effect of back support use on comfort | 6 hour
  The immobilization comfort scale consists of 20 items and 6 statements. The total score is between 20 and 120. Scoring was done before and after back support.

SECONDARY OUTCOMES:
Effect of back support use on pain | 6 hour
  The numbers on the pain scale (VAS) are ranked from 0 to 10 at equal intervals, with pain intensity of 1-3 indicating mild pain; 4-6 indicating moderate pain; and 7-10 indicating severe pain. Scoring was done at 0th hour (before back support), 3rd hour (during back support) and 6th hour (after back support).

CONTACTS AND LOCATIONS:
Locations (1):
- Tunceli State Hospital, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No